CLINICAL TRIAL: NCT02020850
Title: Determining the Normal Toe-Brachial Index in Young Adults
Brief Title: Young Toe-Brachial Index Assessment
Acronym: TBI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Other Study IDs: H13-03144
Record Dates: First submitted 2013-12-19; First posted 2013-12-25 (Estimated); Last update posted 2014-07-04 (Estimated); Status verified 2014-07

CONDITIONS: Diabetes Mellitus; Coronary Artery Disease,; Vascular Diseases
Keywords: Toe-Brachial Index; Ankle-Brachial Index; Systolic blood pressure
MeSH Terms: conditions — Diabetes Mellitus; Coronary Artery Disease; Vascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Toe-Brachial and Ankle-Brachial Index: toe systolic blood pressure, ankle systolic blood pressure, brachial systolic blood pressure test

SUMMARY:
The Toe-Brachial Index (TBI) that has been using in our laboratory is 0.6, but the average value we measured in normal individuals is about 1.0, furthermore, we can not find out the reference of TBI that is currently being used. The purpose of this study is to determine the more accurate value of TBI and Ankle-Brachial Index (ABI). In this study, all participants will be required to fill out a demographic questionnaire before the blood pressures test. All participants will have their toe, ankle and brachial systolic blood pressure measurements to obtain the TBI and ABI.

DETAILED DESCRIPTION:
All participants will fill out a demographic questionnaire that includes:

* Race, gender, age
* Height and weight
* Perceived stress level (potentially measured using Cohen's Perceived Stress scale(PSS))
* Activity level, with description hours per week, cardio versus non-cardio, and intensity (mild, moderate, intense)
* Smoking history, alcohol consumption, caffeine intake, and drug use (recreational, medicine - over - the - counter and prescription, including birth control pills)
* Hand dominance, and leg dominance
* Past medical history - with emphasis on cardiovascular disease (hypertension, cancer, coronary heart disease, diabetes mellitus, high cholesterol, coagulopathies, previous thromboses) as well as renal, adrenal, and thyroid disorders, Raynaud's phenomenon
* Family medical history (cancer, coronary heart disease, diabetes mellitus, high cholesterol)

Participants with known existing diabetes, coronary artery disease, or a history of vascular disease will be included in the study; nevertheless, their results may be analyzed in a separate cohort for comparison against those undiagnosed with the aforementioned condition.

The TBI (Toe - Brachial Index) will be measured by the following procedure.

* The assessment time and room temperature will be recorded
* The participant should lay supine for a minimum of five minutes in a warm and comfortable room
* Select the appropriate cuff for each upper arm and each large toe and separately placed them around the arm and large toe.
* The blood pressure measurements will be performed with photo plethysmography (PPS) and chart recorder. The phototransducer is connected to the PPS, and the digit cuff is connected to an aneroid sphygmomanometer.
* The toe and ipsilateral arm systolic blood pressures will be measured up to three times for accuracy.
* The TBI will be calculated by dividing the averaged toe systolic blood pressure, by the averaged brachial systolic blood pressure.

The ABI (Ankle - Brachial Index) will be measured by the following procedure.

* The blood pressure cuff will be placed proximal to the malleoli and ultrasound gel cover the skin overlying the dorsalis pedis and posterior tibial arteries in the foot.
* The dorsalis pedis and posterior tibial arteries blood pressure will be measured by using hand-held Doppler probe.
* The ankle systolic blood pressure will be taken as the higher pressure of the 2 arteries at the ankle.
* The ABI will be calculated by dividing the ankle systolic blood pressure, by the averaged brachial systolic blood pressure.

The brachial, toe and ankle blood pressures will be measured on the opposite limbs, and the TBI and ABI will be calculated following the protocol outlined above.

ELIGIBILITY:
Inclusion Criteria:

* All students from the University of British Columbia, Faculty of Medicine graduating class of 2017

Exclusion Criteria:

* Students who declined to participate in the study

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants will be recruited from the classes of Faculty of Medicine in the University of British Columbia
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-02; Primary Completion 2014-09 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Toe-Brachial Index | Minimum 5 minutes post participant lying supine
  The toe and ipsilateral brachial systolic blood pressures will be measured on both side of limbs. The participant should be fully-supported, comfortable, warm with arms and legs at heart level.

SECONDARY OUTCOMES:
Ankle-Brachial Index | Minimum 5 minutes post participant lying supine
  The ankle and ipsilateral brachial systolic blood pressures will be measured on both side of limbs. The participant should be fully-supported, comfortable, warm with arms and legs at heart level.

CONTACTS AND LOCATIONS:
Overall Officials: York N Hsiang, MB FRCSC, Principal Investigator — UBC, Division of Vascular Surgery and Vancouver General Hospital
Locations (1):
- Vancouver General Hospital (VGH) - Gordon and Leslie Diamond Health Care Centre, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Quong WL, Fung AT, Yu RY, Hsiang YN. Reassessing the normal toe-brachial index in young healthy adults. J Vasc Surg. 2016 Mar;63(3):652-6. doi: 10.1016/j.jvs.2015.09.019. PMID 26916582